CLINICAL TRIAL: NCT06747169
Title: Efficacy and Safety of PD-1 Inhibitor Combined with Nab-PP Plus Rh-endostatin in Locally Advanced/advanced and Recurrent Metastatic Squamous Non-small Cell Lung Cancer: a Single-arm, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Sintilimab Combined with Nab-PP Plus Rh-endostatin in Locally Advanced/advanced and Recurrent Metastatic Squamous Non-small Cell Lung Cancer: a Single-arm, Multicenter Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jian-Guo Zhou, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Jian-Guo Zhou, MD, PhD, associate professor and associate chief physician, Second Affiliated Hospital of Zunyi Medical University
Organization: Second Affiliated Hospital of Zunyi Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-2024-061
Record Dates: First submitted 2024-12-14; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Squamous Non-Small Cell Lung Cancer SqNSCLC
MeSH Terms: interventions — sintilimab; Albumin-Bound Paclitaxel; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Locally Advanced/Advanced or Recurrent Metastatic Sq-NSCLC (Experimental): This cohort includes patients with locally advanced, advanced, or recurrent metastatic squamous non-small cell lung cancer (Sq-NSCLC).
  Interventions: Drug: Sintilimab, albumin-bound paclitaxel plus platinum agent (Nab-PP), and recombinant human endostatin

INTERVENTIONS:
Drug: Sintilimab, albumin-bound paclitaxel plus platinum agent (Nab-PP), and recombinant human endostatin — All patients were treated with a combination therapy consisting of sintilimab, albumin-bound paclitaxel plus platinum agent (Nab-PP), and recombinant human endostatin. The study is designed to assess the efficacy and safety of this treatment regimen in the specified population.

SUMMARY:
The goal of this single-arm, multi-center phase II clinical study is to evaluate the efficacy and safety of recombinant human endostatin (rh-Endostatin) combined with nab-paclitaxel, platinum-based chemotherapy, and PD-1 inhibitors in patients with locally advanced, advanced, or recurrent metastatic squamous non-small cell lung cancer (NSCLC).

The main questions it aims to answer are:

What is the progression-free survival (PFS) and objective response rate (ORR) of this combination therapy? What is the safety profile, including adverse event (AE) and serious adverse event (SAE) rates? Researchers will compare the treatment effects over time by evaluating tumor responses using RECIST 1.1 criteria and assessing quality of life using the EORTC QLQ-C30 (v3.0) and QLQ-CX24 scales.

Participants will:

Receive 4-6 cycles of rh-Endostatin combined with nab-paclitaxel, platinum-based chemotherapy, and PD-1 inhibitors.

Continue maintenance treatment with rh-Endostatin and PD-1 inhibitors until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must voluntarily participate in the study and provide written informed consent.
2. Age between 18 and 70 years, applicable to both sexes.
3. Histologically or cytologically confirmed advanced or metastatic (Stage IIIB, IIIC, or IV) squamous NSCLC without driver gene mutations.
4. At least one measurable target lesion per RECIST 1.1 criteria, untreated with local therapies (e.g., radiotherapy).
5. ECOG performance status score of 0-1.
6. Expected survival ≥ 3 months.
7. Treatment-naïve patients (no prior systemic anti-tumor therapy, including radiotherapy, chemotherapy, targeted, or immunotherapy), or patients with recurrence ≥ 6 months after adjuvant chemotherapy.
8. Adequate organ function within 7 days prior to treatment:

1）Hematology (without recent blood transfusion): Hemoglobin (HB) ≥ 90 g/L Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelets (PLT) ≥ 80 × 10⁹/L 2）Biochemistry: Total bilirubin (TBIL) ≤ 1.5 × ULN ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN for liver metastases) Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60 mL/min Serum albumin ≥ 35 g/L 3) Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%. 9.Tissue samples required for biomarker analysis (e.g., PD-L1): newly obtained samples are preferred. Archived samples (collected within 2 years prior to enrollment) are acceptable, with 3-5 μm paraffin sections (5-8 slides).

Exclusion Criteria:

1. History of severe hypersensitivity or allergic reactions to humanized antibodies or fusion proteins.
2. Known hypersensitivity to recombinant human endostatin or any component of antibody preparations.
3. Diagnosed with immunodeficiency or receiving systemic corticosteroids or other immunosuppressive therapies within 14 days prior to the first dose of study treatment (physiologic doses of corticosteroids, such as ≤10 mg/day prednisone or equivalent, are allowed).
4. Active, known, or suspected autoimmune diseases (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hypothyroidism). However, patients with Type 1 diabetes, hypothyroidism requiring only hormone replacement, skin conditions not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia), or autoimmune conditions not expected to recur in the absence of external triggers may be included.
5. Pre-existing severe cardiac conditions, including congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina, myocardial infarction, or severe valvular disease.
6. Prior treatment with anti-angiogenic drugs (e.g., bevacizumab, sunitinib, sorafenib, imatinib, famitinib, regorafenib, apatinib, anlotinib).
7. Planned systemic anti-tumor therapy (e.g., cytotoxic therapy) within 4 weeks before randomization or during the study.
8. Active hepatitis B (HBV DNA ≥2000 IU/ml or 10⁴ copies/ml) or active hepatitis C (positive anti-HCV and detectable HCV RNA).
9. Active tuberculosis (TB) infection based on chest X-ray, sputum examination, or clinical assessment. Patients with a history of active TB within the past year, even if treated, are excluded. Patients with a history of TB more than one year ago may participate only if prior anti-TB treatment was deemed appropriate.
10. Symptomatic brain metastases or brain metastases with symptom control <2 months.
11. Major surgical procedures, incisional biopsy, or significant traumatic injuries within 28 days prior to randomization.
12. Tumors invading major blood vessels or with a high risk of vascular invasion and fatal hemorrhage, as determined by investigators.
13. Evidence or history of bleeding diathesis, regardless of severity. Patients with unresolved wounds, ulcers, or fractures, or those experiencing bleeding events ≥CTCAE Grade 3 within 4 weeks prior to randomization are excluded.
14. Venous or arterial thrombotic events (e.g., stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the past 6 months.
15. Any comorbidity that, in the investigator's judgment, pose a significant risk to patient safety or interfere with study completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-17 (Estimated); Primary Completion 2026-12-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the initiation of treatment (Day 1) until the first occurrence of disease progression, death, or the end of the study, whichever came first，up to approximately 5 years.
  PFS refers to the length of time from the start of treatment until the tumor progresses or the patient dies, typically assessed through imaging or clinical evaluation. This endpoint reflects the effectiveness of the treatment in delaying disease progression. PFS is particularly useful in evaluating the clinical efficacy of new drugs or therapies. An extension of PFS is usually considered a sign of effective treatment.

SECONDARY OUTCOMES:
Overall survival（OS） | From the initiation of treatment (Day 1) until death or the end of the study, whichever occurs first, up to approximately 7 years
  OS is defined as the time from the initiation of treatment to the date of death from any cause. If a patient is alive at the end of the study or lost to follow-up, OS will be censored at the last known date of follow-up.
Adverse Events (AE) and Serious Adverse Events (SAE) | From the initiation of treatment (Day 1) until 90 days after the last dose of treatment.
  Safety and tolerability will be assessed by recording the incidence of adverse events (AEs) and serious adverse events (SAEs). The proportion of patients experiencing AEs/SAEs and the proportion of events leading to treatment discontinuation will be recorded and analyzed.
Objective response rate(ORR) | Assessed after every two cycles of treatment (each cycle is 21 days) through study completion, up to 5 years.
  ORR refers to the proportion of patients who achieve either a complete response (CR) or partial response (PR) during treatment. This endpoint reflects the effectiveness of the treatment in controlling the tumor. It is typically assessed through imaging techniques (e.g., CT, MRI) and scored based on RECIST (Response Evaluation Criteria in Solid Tumors) or similar criteria. ORR is a common efficacy endpoint in cancer clinical trials.

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.